CLINICAL TRIAL: NCT04443205
Title: Relevance of Ultrasound Screening for Foetal Macrosomia and Description of Its Management in Champagne-Ardenne
Brief Title: Relevance of Ultrasound Screening for Foetal Macrosomia
Acronym: USmacro
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PO20090
Record Dates: First submitted 2020-06-17; First posted 2020-06-23 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Pregnancy
Keywords: Fetal Macrosomia; Ultrasound; Shoulder Dystocia; induction of labour; Cesarean
MeSH Terms: conditions — Fetal Macrosomia; Shoulder Dystocia | interventions — Electronic Health Records

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- no macrosomy: pregnant women whose child is not macrosomal
  Interventions: Other: Data record
- screened macrosomy: pregnant women whose child is macrosomal and have been screened g using ultrasound during the third trimester of pregnancy
  Interventions: Other: Data record
- no screened macrosomy: pregnant women whose child is macrosomal and havenot been screened g using ultrasound during the third trimester of pregnancy
  Interventions: Other: Data record

INTERVENTIONS:
Other: Data record — Data record

SUMMARY:
Management of fetal macrosomia is based on a suspicion of macrosomia (no certainty before birth). This management is an artificial induction of labour for an earlier delivery and therefore a lower fetal weight gain. Several studies have already shown that ultrasound performed during the third trimester of pregnancy was not a perfect tool for this screening.

DETAILED DESCRIPTION:
The aim of the study is to describe management of women whose child is macrosomal but has not been screened g using ultrasound during the third trimester of pregnancy.

ELIGIBILITY:
Inclusion criteria : Patients (consecutive inclusions) :

Women pregnant Women followed in the gynaecology and obstetrics department of the CHU of Reims, the CHG of Charleville Mézières or the CHG of Chalons en Champagne.

Women for which the delivery is planned in the gynaecology and obstetrics department of the Reims University Hospital, the Charleville Mézières General Hospital or the Chalons en Champagne General Hospital.

Non-inclusion criteria Women without ultrasound dating scan in the first trimester. Women having a contraindication to labour or vaginal delivery Women with a scarred uterus Women having a history of shoulder dystocia or obstetric trauma Women having a history of urinary or fecal incontinence Women having a history of bad birth experience with high psychological impact Women with maternal pathologies (excluding gestational diabetes) Women whose fetus is breech Women with twin pregnancy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Foetal macrosomia | Baseline
  estimated weight above the 90th percentile of the curves of the French College of Fetal Ultrasound during the third trimester ultrasound

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France